CLINICAL TRIAL: NCT03497000
Title: Effects of Optical Coherence Tomography Angiography-guided Photodynamic Therapy in Acute Central Serous Chorioretinopathy
Brief Title: Effects of OCTA-guided PDT in Acute CSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Mingwei Zhao, Head of Ophthalmology, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Peking UPH
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Central Serous Chorioretinopathy; Tomography, Optical Coherence
Keywords: optical coherence tomography angiography; central serous chorioretinopathy; photodynamic therapy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCTA group (Experimental): Patients in this group underwent OCTA-guided half-dose photodynamic therapy.
  Interventions: Procedure: OCTA-guided Photodynamic therapy
- ICGA group (Active Comparator): Patients in this group underwent normal ICGA-guided half dose photodynamic therapy.
  Interventions: Procedure: ICGA-guided Photodynamic therapy

INTERVENTIONS:
Procedure: OCTA-guided Photodynamic therapy — Half-dose photodynamic therapy using verteporfin under the guidance of OCTA
  Arms: OCTA group
Procedure: ICGA-guided Photodynamic therapy — Half-dose photodynamic therapy using verteporfin under the guidance of ICGA
  Arms: ICGA group

SUMMARY:
OCTA-guided PDT is as safe and effective as ICGA-guided PDT in the treatment of acute central serous chorioretinopathy. Or OCTA-guided PDT is more effective than ICGA-guided PDT in the treatment of acute central serous chorioretinopathy, safe as well.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic detachment of the neurosensory retina with a focal leak at the level of the RPE with FA
* Presence of SRF and/or serous pigment epithelial detachment on OCT
* Presence of abnormal dilated choroidal vasculature in ICGA

Exclusion Criteria:

* Patients with other ocular conditions commonly associated with SRF, such as choroidal neovascularization, polypoidal choroidal vasculopathy (PCV), diabetic retinopathy, retinal vascular occlusion, Coat's disease
* Any disease that may affect the quality of imaging (quality of OCTA images < 6), such as cataract, high myopia or nystagmus
* History of ocular surgeries including retinal laser
* Pregnancy
* Any uncontrolled systemic disease
* Any condition rendering patients intolerable to image acquisition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Number of patients with subretinal fluid resolution on OCT after PDT of two groups | 3 months

SECONDARY OUTCOMES:
Number of patients with leakage point resolution on FFA after PDT of two groups | 3 months
Number of recurrent CSC after PDT of two groups | 3 months
BCVA (best corrected visual acuity) at every follow-up of two groups | 1 month, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei Zhao, M.D, Study Director — Peking University People's Hospital
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hu J, Qu J, Li M, Sun G, Piao Z, Liang Z, Yao Y, Sadda S, Zhao M. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY-GUIDED PHOTODYNAMIC THERAPY FOR ACUTE CENTRAL SEROUS CHORIORETINOPATHY. Retina. 2021 Jan 1;41(1):189-198. doi: 10.1097/IAE.0000000000002795. PMID 32343102